CLINICAL TRIAL: NCT04354935
Title: Treatment of Resistant Depression by Repetitive Transcranial Magnetic Stimulation (rTMS) Multicentric Naturalistic Study
Acronym: DSNATUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Noomane Bouaziz, MD, psychiatrist, Centre hospitalier de Ville-Evrard, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10477M-DSNATUR-2020
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: To Evaluate the Effectiveness of Open rTMS
Keywords: rTMS; TMS; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Multicentric Naturalistic Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Method 1 ( iTBS) (Active Comparator): target region: Dorsolateral Prefrontal left Fréquence : 50 Hz Intensity of the stimulation : 120% SM duration : 3 minutes Number of pulses : 600
  Interventions: Device: rTMS basic
- Method 2 (French touch) (Active Comparator): target region : dorsolateral prefrontal cortex right Frequency:1HZ Intensity:120% SM duration : 8 Min 30 Sec Number of plulses : 360
  Interventions: Device: rTMS basic
- Method 3 (FDA) (Active Comparator): target region: Dorsolateral Prefrontal left Fréquence : 10HZ Intensity of the stimulation : 120% SM duration : 37 minutes Number of pulses : 3000
  Interventions: Device: rTMS basic
- Method 4 (ITBS VIIT) (Active Comparator): target region: Dorsolateral Prefrontal left Fréquence : 50HZ Intensity of the stimulation : 90% SM Duration : 9 minutes Number of pulses : 1800
  Interventions: Device: rTMS VIIT
- Method 5 (SNTm) (Active Comparator): Target region: Dorsolateral Prefrontal left Fréquence : 50HZ Intensity of the stimulation : 90% SM Duration : 9 minutes Number of pulses : 1800
  Interventions: Device: rTMS SAINT modified
- Method 6 (SNT) (Active Comparator): Target region: Dorsolateral Prefrontal left Fréquence : 50HZ Intensity of the stimulation : 90% SM Duration : 9 minutes Number of pulses : 1800
  Interventions: Device: rTMS SAINT
- Method 7 (DASH) (Active Comparator): Target region: Dorsolateral Prefrontal left Fréquence : 10HZ Intensity of the stimulation : 120% SM Duration : 18.75 minutes Number of pulses : 3000
  Interventions: Device: rTMS basic

INTERVENTIONS:
Device: rTMS basic — 1 session per day, for 4 or 6 weeks.
  Arms: Method 1 ( iTBS); Method 2 (French touch); Method 3 (FDA); Method 7 (DASH)
Device: rTMS VIIT — 5 sessions per day, for 2 weeks.
  Arms: Method 4 (ITBS VIIT)
Device: rTMS SAINT modified — 8 sessions per day, for 1 week.
  Arms: Method 5 (SNTm)
Device: rTMS SAINT — 10 sessions per day, for 1 week.
  Arms: Method 6 (SNT)

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) for repetitive Transcranial Magnetic Stimulation) is a a recent technique to stimulate the brain in a way that non-invasive, for therapeutic purposes. The first trials of analgesic use of rTMS date back to about 15 years ago. years and clinical use has now entered the practice of some specialized centers. Used at a frequency less than or equal to 1 Hertz (Hz; a stimulation per second), it is called bass rTMS. frequency and results in inhibition of cortical excitability at the level of the stimulated area. Conversely, a stimulation with a frequency higher than 5 Hz, called high-frequency rTMS, will have an excitatory effect on the targeted neurons. In addition to its local effects at the stimulation site, rTMS can also have effects on distance on regions other than those directly targeted. The impact of this treatment would be the local modulation of the cerebral plasticity and also act on the anatomical connectivity and functional brain function in both healthy subjects and those who are patients with psychiatric disorders

DETAILED DESCRIPTION:
Main objective :

To show the effectiveness of rTMS carried out in open on the symptoms of depression resistant in common practice between the Baseline and the end of the initial treatment (between 1 and 6 weeks).

Secondary Objectives

Evaluate the tolerance of the rTMS carried out in open on the symptoms of depression resistant in common practice between the Baseline and the end of the initial cure (between 1 and 6 weeks)

Evaluate the impact of this treatment on :

* The response rate
* The remission rate
* Quality of life To assess the correlation between personality dimensions and depression.

The criteria main evaluation :

The evolution of the HDRS-17 score (Hamilton depression scale, 17 items) between the Baseline and the end of the initial treatment (1 to 6 weeks)

The evaluation criteria secondary :

* Responder patient rate (defined as a 50% decrease in the rate of

  % of HDRS score)
* Rate of patients in remission (defined by HDRS score<8)
* Evolution of the EQ5D quality of life score between Baseline and end of the initial treatment (between 1 and 6 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Presenting a depressive episode characterized as resistant according to the DSM 5 criteria
* resistance is characterized by: non-response to at least two different antidepressants prescribed at effective doses for a duration greater than or equal to 6 weeks.
* Patient who agrees to participate in the study and who has signed an informed consent.
* Patient fluent in French
* Affiliation to a social security scheme.
* Women of childbearing age must be on contraception

Exclusion Criteria:

* Presenting a contraindication to TMS: intrafemale foreign body cranial, unstable epilepsy, cochlear implant, pacemaker, pregnancy
* Presence of a psychotic disorder
* Presence of an unstable medical condition
* Presence of schizophrenia or persistent delusional disorder
* Persons under guardianship, curatorship and safeguarding of justice.
* Pregnant women,
* Woman of childbearing age without effective contraception
* Breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
measure the evolution of the HDRS-17 score | an average of 1 year
  The evolution of the HDRS-17 score (Hamilton depression scale, 17 items) between the Baseline and the end of the initial 4 to 6 week treatment course

SECONDARY OUTCOMES:
Rate of responding patients | an average of 1 year
  Rate of responder patients (defined by a 50% decrease in HDRS score)
Rate of patients in remission | an average of 1 year
  defined by HDRS score<8
Evolution of the quality of life score | an average of 1 year
  EQ5D between Baseline and the end of the initial treatment between 4 and 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Youcef Bencherif, Neuilly-sur-Marne
  - Unité de recherche clinique, Neuilly-sur-Marne, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No